CLINICAL TRIAL: NCT05754177
Title: Evaluating the Safety and Efficacy of a Probiotic on IBS Symptom Severity in Adults With Diarrhoea-predominant Irritable Bowel Syndrome
Brief Title: Safety and Efficacy of a Probiotic Supplement in IBS-D
Acronym: IBIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Vizera d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ADM/CTB2022TN102
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome With Diarrhea; Irritable Bowel Syndrome
Keywords: IBS; Probiotic; Irritable Bowel Syndrome; GI microbiome; Bifidobacterium
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Arm receiving investigation product (probiotic)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Arm receiving placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants in this arm will receive a daily dose of 1x10^10 Colony Forming Unit (CFU) of a single strain probiotic (live bacteria), administered orally by 1 capsule a day, for 84 days
  Arms: Probiotic
Other: Placebo — Participants in this arm will receive an equivalent placebo for 84 days.
  Arms: Placebo

SUMMARY:
This study aims to assess the safety and efficacy of a single probiotic strain on symptom severity in adults with diarrhea-predominant Irritable Bowel Syndrome (IBS-D).

DETAILED DESCRIPTION:
This is a double-blind, randomised, placebo-controlled trial designed to assess the safety and efficacy of a single probiotic strain on symptom severity in adults with IBS-D, when consumed orally in capsule form once daily for 84 days. Volunteers will be screened in order to identify up to 134 participants meeting ROME IV criteria for IBS-D. The study will involve 5 visits over a total of 105 days [visit 1: screening, commencement of run in period (-21 to -14 days), visit 2: baseline/ randomisation (day 0), visits 3 and 4: intervention period (day 28 ± 2, day 56 ± 2), visit 5: end of study (day 84± 2)]. Participants will fill in daily and weekly eDiaries, and questionnaires will be administered at study visits. Faecal samples will be collected on visits 2 and 5.

ELIGIBILITY:
Inclusion criteria

* Males and females aged ≥18 to ≤ 65 years.
* Participants diagnosed with diarrhoea-predominant irritable bowel syndrome (IBS-D) as per ROME IV criteria:

  i) Recurrent abdominal pain on average at least one day/week in the last three months, associated with two or more of the following criteria:
  * Related to defecation
  * Associated with a change in stool frequency (increase/decrease in frequency).
  * Associated with a change in the form (appearance) of stool. ii) History of abnormal bowel movements predominantly diarrhoea (>25% of bowel movements categorised as stool form type 6 or 7 (diarrhoea) and <25% as stool form type 1 or 2 (constipation) on BSFS).
* Participants with an IBS-SSS score ≥ 175.
* Participants who test negative for COVID-19 by Rapid Antigen Test Device.
* Participants who did not change their diet within three months before the screening day and are willing to sustain that diet during the study.
* Participants who can comply and perform the procedures as per the protocol (consumption of study products, biological sample collection procedures, and study visit schedule).
* Participants who are literate enough to understand the purpose of the study and their rights.
* Participants who are able to give written informed consent and are willing to participate in the study.

Exclusion criteria

* Participants who score ≥ 40 in either the 'state' or 'trait' section of the STAI-AD questionnaire (both sections to be assessed).
* Participants diagnosed with Coeliac Disease.
* Lactose intolerant participants unless on a strict lactose free diet for at least three months before screening day with persistent symptoms of IBS-D.
* Participants with a body mass index (BMI) ≥ 30 kg/m2.
* Presence of uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 140 mm Hg and/or diastolic blood pressure (DBP) ≥ 90 mm Hg.
* Participants with a history of intake of antibiotics (Rifaximin, metronidazole, or any other), other probiotics, prebiotics, synbiotics, food supplements with iron or calcium, peppermint oil, acid sequestrants (cholestyramine, Bile colestipol), introduced/active low FODMAP diet, and histamine H2-receptor antagonists/H2 blockers within six weeks prior to the screening day.
* Participants with a history of daily intake of antidepressants (Tricyclic antidepressants, Selective serotonin reuptake inhibitors (SSRIs), and Selective serotonin-norepinephrine reuptake Inhibitors (SSNRIs)), clonidine, otilonium bromide, asimadoline, eluxadoline, diphenoxylate, antispasmodics including mebeverine and pinnaverium and anticholinergics within two weeks prior to the screening day.
* Participants with a history of bariatric surgery or surgical resection of the stomach, small intestine, or large intestine.
* Participants with a history of gastrointestinal-related abdominal surgery other than hernia repair.
* Participants with a history of or complications from inflammatory bowel disease (Crohn's disease or ulcerative colitis) and ischemic colitis.
* Participants showing signs of bile acid malabsorption (BAM), as evident from the history of green colour or foul odour of the stool during the last month.
* Participants with a history of or complications from GI malignant tumours.
* Participants with a history of or complications from other malignant tumours in the last 5 years.
* History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's endpoints.
* Participation in other clinical studies in the last 90 days prior to screening day.
* Active smokers or using any form of smokeless tobacco.
* Participants with substance abuse problems (within two years) defined as:

  * Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
  * High-risk drinking as defined by the consumption of four or more alcohol-containing beverages on any day or eight or more alcohol-containing beverages per week for women and five or more alcohol-containing beverages on any day or 15 or more alcohol-containing beverages per week for men.
* Participants having clinically significant illnesses of cardiovascular, endocrine, immune, respiratory, hepato-biliary, kidney and urinary, haematological, musculoskeletal system and/or any inflammatory disorder and other gastrointestinal diseases.
* Participants with active human immunodeficiency virus (HIV) or hepatitis A, B or C infection.
* Female participants being pregnant, breastfeeding or planning pregnancy in the course of the study.
* Any condition that could, in the opinion of the Investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in total irritable bowel syndrome symptom severity score (IBS-SSS) | Day 0, Day 28, Day 58 and Day 84
  Change in IBS-SSS totals score (max 500 points) from baseline to day 28, day 58 and day 84, where higher scores mean worse outcomes

SECONDARY OUTCOMES:
Percentage of population achieving a normal stool consistency | Day 0, Day 28, Day 58 and Day 84
  Percentage of the population achieving normal stool consistency, defined as over 75% of total bowel movements classified as stool form type 3, 4, and 5 on Bristol Stool Form Scale (BSFS) (BSFS range: 1-7, lower scores mean constipation, higher scores mean diarrhea). Weekly percentage at baseline compared to weekly percentage at day 28, 58 and 84.
Percentage of population without diarrhea | Weekly
  Percentage of the population where less than 25% of bowel movements are diarrhea, defined as stool form type 6 or 7 on the Bristol Stool Form Scale (BSFS) (BSFS range: 1-7, lower scores mean constipation, higher scores mean diarrhea). Weekly percentage calculated throughout study and compared to baseline weekly percentage.
Change in Irritable Bowel Syndrome Quality of Life (IBS-QOL) score | Day 0, Day 28, Day 58 and Day 84
  Change in quality of life, assessed by change in the IBS-QOL total score (max 100 points) between baseline and day 28, day 58 and day 84, where higher scores mean better quality of life
Change in State-Trait Anxiety Inventory for Adults (STAI-AD) score | Day 0, Day 28, Day 58 and Day 84
  Mental health as assessed by change in STAI-AD S-anxiety subscale score (max: 80), between baseline and day 28, 58 and 84, where higher scores mean more severe anxiety symptoms
Gut microbiome compositional changes | Day 0, Day 84
  Change in gut microbiome composition, as assessed by shotgun sequencing of faecal samples, between baseline and study end (day 84)
Use of Rescue Medication | Day 0, Day 84
  Comparison in total cumulative use of rescue medications between the two study arms at study end (day 84)

OTHER OUTCOMES:
Adverse Events | Day 0, Day 84
  Comparison in the total number of adverse events/serious adverse events occurred during the study, from baseline to study end (day 84), between the two study arms
Stool Biochemistry | Day 0, Day 84
  Change in stool faecal biochemistry between baseline and study end (day 84) between the two study arms
Proton Pump Inhibitor Use | Day 0, Day 84
  Subpopulation analysis: participants taking proton pump inhibitors (PPIs) and participants not taking PPIs compared to placebo at study end

CONTACTS AND LOCATIONS:
Locations (1):
- Vizera, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No